CLINICAL TRIAL: NCT01915043
Title: Improving Adherence Healthy Lifestyle With a Smartphone Application Based After Surgery in Cancer Patients
Acronym: APPCOMCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: FCCSS_UMA-02-13
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2017-03

CONDITIONS: Secondary Prevention
Keywords: lymphedema, prevention, ehealth, cancer
MeSH Terms: conditions — Lymphedema; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- health education for lymphedema prevention (Active Comparator): health education for lymphedema prevention
  Interventions: Other: health education for lymphedema prevention
- application smartphone-based group (Experimental): Health education plus Smartphone-based application sample will have a reminder to do education everyday where patients will have to select if they have done or they haven´t done compliance
  Interventions: Other: health education for lymphedema prevention

INTERVENTIONS:
Other: health education for lymphedema prevention — All subjects received a multimodal intervention consist in a multimodal program with an educational approach

SUMMARY:
Background: The cancer-related lymphedema (BCRL) is the abnormal accumulation of fluid in the lymphatic system and can develop immediately after surgery / radiotherapy of breast cancer, or may appear months later. In the literature there are numerous educational recommendations to avoid the appearance BCRL, but there is a lack of adherence to these recommendations. With the increase of mobile technologies among adults, the mobile devices can be an effective method to meet their education.

Objective: To determine the effectiveness of therapeutic adherence a brief educational intervention through a smartphone-based application in the prevention of lymphedema in women with mastectomies.

Method: 100 women survivors of breast cancer will be randomized to a group that will receive lymphedema prevention education and an app specific for better adhesion compared to the control group will receive education only. They will be monitored for 28 weeks by specific measures of lymphedema onset, volume and perimeter arm and hand strength lymphedema disability questionnaire and other measures of fatigue, quality of life and mood related to cancer.

Discussion: The lack of adherence to health education is the main cause of failure in maintaining these brief educational interventions, whether the program is beneficial, it could be successfully implemented in clinical practice.

ELIGIBILITY:
Women diagnosed with breast cancer, including the Via Clinic (11) breast cancer at the Hospital Costa del Sol, Marbella, Spain.

Inclusion criteria :

* be over 18 years
* with own smartphone telephony server and mobile internet.

Exclusion criteria :

* reading problems, psychological problems, who can not read Spanish
* unwilling to participate in the study.

It also takes into account the severity of the disease, dividing criteria, conservative surgery, mastectomy, with or without lymphadenectomy, sentinel node.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
volume and perimeter arm | baseline and 18 weeks
  Water Displacement (volume) Is performed by the water displacement method, a volumeter to reference point 16 cm proximal to the olecranon, with a Tª of 21ºC. The upper limit is 65% of the distance from the olecranon to the acromion.
  Circumferential Measurement (Perimeter) The patient should be seated both arms on a table, shoulder in neutral rotation and in flexion of 45º, forearm in maximun supination, is measured at intervals of 5 cm along both arms, using elbow crease as starting point.

SECONDARY OUTCOMES:
hand strength | baseline; 18 and 28 weeks
  It´s a standardized method to evaluate the hand strengh and it´s relation to the function of the upper extremity. Is done with a Jamar hydraulic hand dynamometer, has 5 fixed grip posititons.
Quality of Life Breast CAncer QLQ-BR23 questionnaire | baseline; 18 and 28 weeks
  The QLQ-BR23 consist of 23 items, is divided in dimennsions as body image, sexuality, future perspective and side-effects to different treatment modalities such as surgery, chemotherapy or radiotherapy.
Cancer related fatigue questionnaire | baseline; 18 and 28 weeks
  Quick-Piper scale, self- administered, a 15 items. Consists of 4 subjetive dimensions. Offers the important advantage of brevity.
volume and periemter arm | changes from 18 to 28 weeks
  Water Displacement (volume) Is performed by the water displacement method, a volumeter to reference point 16 cm proximal to the olecranon, with a Tª of 21ºC. The upper limit is 65% of the distance from the olecranon to the acromion.
  Circumferential Measurement (Perimeter) The patient should be seated both arms on a table, shoulder in neutral rotation and in flexion of 45º, forearm in maximun supination, is measured at intervals of 5 cm along both arms, using elbow crease as starting point.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Study Director — University of Malaga
Locations (1):
- Hospital Costa del Sol, Marbella, Malaga, Spain